CLINICAL TRIAL: NCT06019988
Title: Early Point-of-Service SBDOH Screening in Breast Cancer
Brief Title: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening and Enhanced Navigation on Care Delivery for Patients With Breast Cancer
Acronym: Breast_SBDOH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Oluwadamilola Fayanju, MD, MA, MPHS, FACS, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19122
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Social Determinants of Health (SDOH)
Keywords: Social and behavioral determinants of health; SDOH; SBDOH; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: All enrolled patients will initially receive one of three screening tools (The Accountable Health Communities Health-Related Social Needs Screening Tool [AHC-HRSN], Health Leads Social Screening Tool, or National Comprehensive Care Network Distress Thermometer and Problem List [NCCN DT+PL]) via the MyPennMedicine patient portal and be given 48 hours to respond. Those patients who do not respond will be randomized to one of two intervention arms, each of which is an alternative modality to receive and respond to the assigned screening tool: a bidirectional text-based conversational agent (chatbot) or interactive voice response system administered by phone.
  There exists three instrument arms (AHC-HRSN, Health Leads, and NCCN DT+PL) and two modality arms (chatbot and IVR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- The Accountable Health Communities Health-Related Social Needs Screening Tool (AHC-HRSN) (Other): Patients will be randomized to receive one of three social needs screening instruments. The AHC-HRSN is a 10-item tool developed by the Centers for Medicare and Medicaid Services to assess patient needs in 5 core domains, including housing instability, food insecurity, transportation problems, utility help needs, and interpersonal safety, with eight supplemental domains to collect information about financial strain, employment, family and community support, education, physical activity, substance abuse, mental health, and disabilities. The AHC-HRSN tool is designed to help physicians identify unmet needs and refer affected patients to appropriate community services.
  Interventions: Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening
- Health Leads Social Screening Tool (Other): Patients will be randomized to receive one of three social needs screening instruments. Health Leads is an 8-item survey with yes/no responses, which screens for food insecurity, utility needs, housing instability, childcare, financial resource strain, transportation challenges, education, and social isolation.
  Interventions: Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening
- National Comprehensive Care Network (NCCN) Distress Thermometer and Problem List (DT + PL) (Other): Patients will be randomized to receive one of three social needs screening instruments. The NCCN Distress thermometer is a single-item tool designed to measure patients' current level of distress. Patients are asked to rate their distress using a 10-point Likert scale, where 0=no distress and 10=extreme distress. The Problem List (PL) helps physicians identify the sources of patients' distress and direct patients to appropriate support services. The NCCN DT+PL is a widely used, validated tool for evaluating distress in patients diagnosed with or receiving treatment for cancer.
  Interventions: Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening
- Chatbot (Other): Patients who do not respond to the survey within 48 hours of being first administered via MyPennMedicine will be sent the same survey via one of two modality arms. The chatbot is a bidirectional text-based conversational agent administered via WaytoHealth. Patients will again have 48 hours to respond via chatbot.
  Interventions: Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening
- Interactive Voice Response (IVR) System (Other): Patients who do not respond to the survey within 48 hours of being first administered via MyPennMedicine will be sent the same survey via one of two modality arms. The interactive voice response (IVR) system is administered via phone through WaytoHealth. Patients will be called over the phone and will receive the screening tool through IVR. Patients will again have 48 hours to respond via IVR.
  Interventions: Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening

INTERVENTIONS:
Other: Early Point-of-Service Social and Behavioral Determinants of Health (SBDOH) Screening — All patients who participate in the trial will receive one of three social and behavioral determinants of health (SBDOH) screening instruments (AHC-HRSN, Health Leads, or NCCN DT + PL). Any patients who do not complete the screening within 48 hours of its administration will be randomized to receive the same screening via one of two modality arms (Chatbot or IVR System)

SUMMARY:
The overarching goal of this project is to optimize the collection of social and behavioral determinants of health (SBDOH) for patients with a pathological diagnosis of breast cancer at Penn Medicine. The investigators will measure rates of SBDOH data collection by modality and rates of referral to and uptake of social support services, time to evaluation, staff time, acceptability, patient-centered communication, medical mistrust, and clinician acceptability.

DETAILED DESCRIPTION:
The investigators will conduct a patient-level, pragmatic opt-out trial to test implementation of a comprehensive, tech-enabled platform for administration of a validated SBDOH screening tool in contrast to the current practice of unstructured social history collection at this institution.

For internally referred patients, study coordinators - who are functioning as patient navigators - will facilitate a warm handoff from radiology to the New Patient Office as well as study introduction and enrollment. If patients do not wish to have a warm handoff call with a new-patient coordinator (NPC) in the NPO who will schedule the patient's consult with a surgeon and/or oncologist, or if patients are diagnosed external to Penn Medicine, the patient coordinator will follow up directly with the patient to facilitate communication and enrollment within 24 hours of diagnosis.

All patients who do not opt out will be part of the analytic cohort and randomized to one of three screening assessment tools:

1. Accountable Health Communities Health-Related Social Needs Screening Tool (AHC-HSRN);
2. Health Leads Social Needs Screening Toolkit (Health Leads);
3. National Comprehensive Cancer Network (NCCN) Distress Thermometer + Problem List (NCCN DT+PL).

   . The initial request for completion will be administered via the institutional EHR's Epic-based patient portal. Patients will have 48 hours to respond and will receive 2 reminders via a MyPennMedicine message (MPM), through which a patient can also indicate a desire to opt-out if they wish.

   Patients who do not respond and remain enrolled will be randomized to either a bidirectional text-based conversational agent (i.e., "chatbot") or interactive voice response (IVR) system administered by phone. Through the first arm, patients will engage with the screening tool through an interactive two-way text messaging chatbot through WaytoHealth©. Through the second arm, patients will be called over the phone and will receive the screening tool through interactive voice recognition. Patients will again have 48 hours to respond and will receive 2 reminders via the modality to which they have been newly randomized. Patients have the opportunity to opt out through either modality and discontinue study.

   Patients who have not completed the screen via any modality by the time of their first surgical consult at Penn after diagnosis, will be provided the opportunity to complete it electronically though a tablet at the clinic appointment. At any point, patients who report challenges with particular SBDOH domains can be referred prior to initial surgical consultation to Social Services at Abramson Cancer Center.

   Approximately 6 months following diagnosis and initial completion in the study trial (Activity 1), a subset of patients (identified via deviant sampling) will be invited to participate in semi-structured interviews (Activity 2) through which mechanisms contributing to the effectiveness of the SBDOH data collection platform will be evaluated. Additionally, clinicians or clinical leaders will be invited to participate in semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

Based on available EHR data, patients will be eligible for Activities 1 and 2 if they:

* Are referred to one of the following locations for surgical consult following a new diagnosis of operable (Stage 0-III) breast cancer: the Hospital of the University of Pennsylvania (HUP), Penn Presbyterian Medical Center (PPMC), Pennsylvania Hospital (PAH), and Penn Medicine Radnor
* Are female
* Are 18 years of age or older, and
* Are able to read and speak English or Spanish

Clinicians and clinical leaders will be eligible for participation in Activity 2 if they:

* Presently work as a clinician or clinical leader in breast surgery or oncology
* Access PennChart as an aspect of their clinical duties
* Are 18 years of age or older
* Are able to read and speak English or Spanish

Exclusion Criteria:

Based on available EHR data, patients will be ineligible if they:

* Are listed as not wanting to be contacted or solicited for research;
* Have known metastatic disease at time of enrollment; and/or
* Do not otherwise meet all of the enrollment criteria

Clinicians and clinical leaders will be ineligible for participation in Activity 2 if they:

* Are not presently engaged in clinical duties or
* Do not otherwise meet all of the enrollment criteria

This study will not exclude men or nonbinary people who may be diagnosed with breast cancer, but investigators anticipate the sample size for these characteristics will be too small to support meaningful analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Rates of SBDOH screen completion prior to initial surgical consult | 1 year
  Rates of SBDOH screen completion prior to initial surgical consult will be first compared by instrument (Accountable Health Communities Health-Related Social Needs Screening Tool [AHC-HRSN], Health Leads Social Needs Screening Toolkit [Health Leads], National Comprehensive Cancer Network Distress Thermometer and Problem List [NCCN DT + PL]). Only the NCCN DT employs a 10-point Likert scale, where 0 = no distress and 10 = extreme distress. Among patients who do not respond to initial screening administration and who then receive the screening via either chatbot or IVR, rates of SBDOH screen completion will be compared by modality.

SECONDARY OUTCOMES:
Time from biopsy to initial surgical consult | 1 years
  Time to evaluation (TTE) will be compared first by instrument (Accountable Health Communities Health-Related Social Needs Screening Tool [AHC-HRSN], Health Leads Social Needs Screening Toolkit [Health Leads], National Comprehensive Cancer Network Distress Thermometer and Problem List [NCCN DT + PL]). Only the NCCN DT employs a 10-point Likert scale, where 0 = no distress and 10 = extreme distress. Among patients who do not respond to initial screening administration and who then receive the screening via either chatbot or IVR, rates of SBDOH screen completion will be compared by modality.
Identify factors associated with rates of post-diagnosis, pre-consultation SBDOH screen completion | 6 months
  Factors associated with rates of SBDOH screen completion across all instruments (AHC-HRSN, Health Leads, and NCCN DT + PL) and modalities will be assessed via individual semi-structured qualitative interviews with patients who participate in Activity 1 as well as clinicians or clinical leaders.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwadamilola Fayanju, MD, Principal Investigator — University of Pennsylvania Division of Breast Surgery
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Reddy KP, Mirpuri S, Berkowitz CL, de Jesus EM, Hulse SB, Lewandowski JT, Coughlin KQ, Burwell ML, Evans R, Galetta J, Rivera Sanchez S, Buckingham TL, Livingstone V, McCarthy AM, Gabriel PE, Edmonds CE, Cadet TJ, Fayanju OM. Implementing social and behavioral determinants of health data collection: insights from a pragmatic trial. JNCI Cancer Spectr. 2025 Apr 30;9(3):pkaf040. doi: 10.1093/jncics/pkaf040. PMID 40408149